CLINICAL TRIAL: NCT03634982
Title: A Phase 1, Open-Label, Multicenter, Dose-Escalation Study of RMC-4630 Monotherapy in Adult Participants With Relapsed/Refractory Solid Tumors
Brief Title: Dose Escalation of RMC-4630 Monotherapy in Relapsed/Refractory Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Revolution Medicines, Inc. (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-4630-01
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumors
Keywords: SHP2; PTPN11; NSCLC; EGFR; KRAS G12; BRAF Class 3; NF1 LOF; advanced solid tumor; advanced solid malignancies; melanoma; skin cancer; ovarian cancer; endometrium/uterus cancer; bladder cancer; cervical cancer; Carcinoma, Non-Small-Cell Lung; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Esophageal Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Neoplasms, Glandular and Epithelial; Gastrointestinal Neoplasms; Digestive System Neoplasms; Head and Neck Neoplasms; Digestive System Diseases; Esophageal Diseases; Gastrointestinal Diseases
MeSH Terms: conditions — Noonan Syndrome; Melanoma; Skin Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Esophageal Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Neoplasms, Glandular and Epithelial; Gastrointestinal Neoplasms; Digestive System Neoplasms; Head and Neck Neoplasms; Digestive System Diseases; Esophageal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RMC-4630 (Experimental): RMC-4630 for oral administration
  Interventions: Drug: RMC-4630

INTERVENTIONS:
Drug: RMC-4630 — RMC-4630 for oral administration

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) profiles of escalating doses of RMC-4630 monotherapy in adult participants with relapsed/refractory solid tumors and to identify the recommended Phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1 study of oral RMC-4630 monotherapy in participants with advanced relapsed or refractory solid tumors. The study will include 2 components: 1) a Dose-Escalation Component for participants with relapsed or refractory solid tumors and 2) a Dose-Expansion Component for participants with relapsed or refractory solid tumors harboring certain specific mutations/rearrangements that result in hyperactivation of the RAS-MAPK pathway. Participants will be treated until disease progression per RECIST v1.1, unacceptable toxicity, or other criteria for withdrawal are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) ≥18 years of age
* Participants who have advanced solid tumors that have failed, are intolerant to, or are considered ineligible for standard of care anticancer treatments including approved drugs for oncogenic drivers in their tumor type
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participants in the Dose-Expansion Component must have one of the following genotypic aberrations: KRAS amplifications, KRASG12C (NSCLC), BRAF Class 3, or NF1 LOF (NSCLC and gynecological cancers) mutations
* Adequate hematologic, hepatic and renal function
* Participant able to understand and voluntarily sign the informed consent form (ICF) and able to comply with the study visit schedule and other protocol requirements.
* Participants willing to agree to not father a child/become pregnant and comply with effective contraception criteria

Exclusion Criteria:

* Known or suspected leptomeningeal or brain metastases or spinal cord compression
* Primary central nervous system (CNS) tumors
* Clinically significant cardiac disease
* Active, clinically significant interstitial lung disease or pneumonitis
* History or current evidence of retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vein occlusion (RVO), or predisposing factors to RPED or RVO
* Known HIV infection
* Active/chronic hepatitis B or C infection
* Any other unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a participant, impact their expected survival through the end of the study participation, and/or impact their ability to comply with the protocol prior/concomitant therapy
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | up to 3 years
  Incidence, nature, and severity of treatment-emergent AEs and serious AEs, including incidence and severity of findings in laboratory values and vital signs for RMC-4630 monotherapy
Number of participants with dose limiting toxicities (DLTs) | 28 days
  Incidence and nature of DLTs with RMC-4630 monotherapy

SECONDARY OUTCOMES:
Cmax | up to 3 years
  Peak plasma concentration of RMC-4630
Tmax | up to 3 years
  Time to achieve peak plasma concentration of RMC-4630
Area Under the Curve (AUC) | up to 3 years
  Area under the plasma concentration time curve of RMC-4630
t1/2 | up to 3 years
  Elimination half-life of RMC-4630
Accumulation Ratio | up to 3 years
  Ratio of accumulation of RMC-4630 from a single dose to steady state with repeated dosing
Overall Response Rate (ORR) | up to 3 years
  Overall response rate of RMC-4630 per RECIST v1.1
Duration of Response (DOR) | up to 3 years
  Duration of response of RMC-4630 per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (12):
- United States (12):
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - UC Irvine - Chao Family Comprehensive Cancer Center, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sarah Cannon Research Institute - Florida Cancer Specialists, Sarasota, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of Texas at Austin - Dell Medical School, Austin, Texas

IPD SHARING:
Plan to Share IPD: No